CLINICAL TRIAL: NCT06166420
Title: Offering Home-based Versus Hospital-based HPV Counseling and Testing for Cervical Cancer Screening in Rural West Region of Cameroon: a Randomised Cluster Trial
Brief Title: Home-based Cervical Cancer Screening Project
Acronym: CASAHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Patrick Petignat (Other)
Collaborators: Dschang District Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Patrick Petignat, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: N°2022/10/1494/CE/CNERSH/SP
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; human papillomavirus; screening; home-based
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Two arms randomised controlled cluster trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home-based (Experimental): A team made up of a Community Health Worker (CHW) and a nurse will do door-to-door sensitization and propose to eligible women to undergo HPV self-sampling test at home. Samples collected will be taken by the nurse to the hospital for HPV testing . Participants will receive a phone call: disclosure of the HPV test's result will be by phone call for HPV-negative participants; HPV-positive participants will be invited to the hospital for disclosure of their results. At the hospital, HP-positive participants will undergo visual assessment of their cervix and treatment if needed.
  Interventions: Other: Experimental
- hospital-based (Active Comparator): Community Health Worker (CHW) will do door-to-door sensitization and invite eligible women to attend cervical cancer screening at District Hospital Dschang. At the hospital they will do HPV self-sampling test. HPV-negative women will be advised to repeat the test after 5 years while HPV positive women will undergo visual assessment of the cervix with acetic acid and lugol (VIA/VILI) and treatment if needed.
  Interventions: Other: Active comparator

INTERVENTIONS:
Other: Experimental — Counseling on cervical cancer screening followed by home-based HPV self-sampling test proposal.
  Arms: home-based
Other: Active comparator — Counseling on cervical cancer screening followed invitation to screen at Dschang District Hospital.
  Arms: hospital-based

SUMMARY:
Cervical cancer is a public health problem in Cameroon.In 2020, the country had a crude incidence of 20.2 per 100 000 women for an incidence to mortality ratio of 0.65. As for now, the country does not have a national screening program to combat the disease. Only 6% of cameroonian women have once been screened for cervical cancer. In order to increase screening uptake so as to reach 70% recommended by the World Health Organization (WHO), a home-based cervical cancer screening approach is proposed. The objective of our study is to compare two recruitment strategies for cervical cancer screening in rural Cameroon.

DETAILED DESCRIPTION:
In 2018, a 5 years cervical cancer screening project called: "Promoting Comprehensive Cervical Cancer Prevention and Better Women's Health in Low- and Medium Resource Settings in the Health District of Dschang" was launched in the West Region of Cameroon. The study aimed at screening 2000 women per year following screen-triage-treatment as recommended by WHO in a 3T approach: Test with HPV self-sampling test, Triage by visual assessement of the cervix with acetic acid and lugol (VIA/VILI), Treatment with thermal ablation. Despite sensitization using communication information channels, uptake of the screening was below the target. In order to increase uptake of the screening, this study proposes a home-based strategy using Community Health Workers (CHW). Community Health Workers (CHW) are lay members of the community who carry out health promotion activities after training. In a randomised controlled cluster trial, two recruitment strategies for cervical cancer screening will be compared: in one arm a team made up of a CHW and a nurse will do door-to-door sensitization and propose home-based HPV self-sampling test to eligible women and in the other arm CHW will do door-to-door sensitization and issue invitation cards to eligible women for hospital-based HPV self-sampling test. This study is nested in ongoing cervical cancer screening project.

Primary objective: To compare completeness of full screening between two different recruitment strategies in rural area: counselling and home-based HPV self-sampling test versus counselling and hospital-based HPV self-sampling test.

Secondary objectives:

* To determine the proportion of women who will carry out an HPV self-sampling test in both strategies within 3 months of sensitization.
* To determine the proportion of HPV positive women who will undergo VIA/VILI in both arms within 3 months.
* To assess the acceptability of home self-sampling HPV test and perception of single versus 2 visits approaches.
* To determine predictors of non-adherence to care-seeking for HPV positive women.
* To determine the number of pre-cancers and/or cancers diagnosed in both arms and their treatment.
* To calculate the economic cost of both strategies.

Mixed method design, quantitative and qualitative informations will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30-49 years
* Ability to understand study procedures and accepting voluntarily to participate by signing an informed consent form (ICF).

Non-inclusion criteria:

* Pregnancy at the time of screening
* History of cervical cancer screening by HPV test of less than 5 years (for HIV-negative women) or less than 3 years (for HIV positive women).
* Intra-vaginal treatment

Exclusion Criteria:

* Symptoms of cervical cancer (e.g. metrorrhagia, known pelvic mass)
* Severe pre-existing medical conditions (e.g. advanced cancer, terminal renal failure)
* Women who are not able to comply with the study protocol.
* Previous hysterectomy
* Known cervical cancer

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 2079 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants who will complete full screening (HPV test +/- VIA/VILI +/- treatment when necessary) in both arms within 3 months of sensitization | 3 months
  The number and percentage of participants who will do an HPV self test+/- VIA/VILI+/- treatment par study arm

SECONDARY OUTCOMES:
Number and percentage of women who will do an HPV test within 3 months of sensitization per study arm | 3 months from sensitization
  The number and percentage of participants who will do an HPV test in each arm of the study.
Number and percentage of participants once tested HPVpositive who will link to the pelvic exam for visual assessment and treatment (if needed) within 3 months. | 3 months from HPV self sample collection
  The number and percentage of participants once tested HPV positive who link to the hospital for visual assessment of the cervix and treatment if needed.
Identify barriers and enablers to the home-HPV self-sampling test. | 4 months
  Factors that prevent and motivate women to participate to a home-based HPV self-test.
Identify barriers and enablers of linkage to VIA for HPV positive women | 4 months
  Factors that prevent and motivate participants who did a home-based HPV self-test to link to the hospital for visual assesment of the cervix using acetic acid and lugol (VIA/VILI).
Number of pre-cancers and/or cancers diagnosed in each study arm. | 2 years
  The number of pre-cancers and cancers diagnosed per study arm.
Cost of each screening strategy. | 2 years
  The cost of each strategy and make a cost-effectiveness analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Petignat, Pr, Principal Investigator — University Hospital, Geneva
Locations (1):
- Dschang District Hospital, Dschang, Menoua, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be shared upon reasonable request at the end of the study period.

REFERENCES:
- [Derived] Moukam AMD, Salah N, Tankeu Happi GW, Metchehe LDD, Makajio SL, Wisniak A, Sormani J, Kenfack B, Vassilakos P, Socpa A, Petignat P, Schmidt NC. Acceptability of home-based HPV self-sampling for cervical cancer screening among users and providers in the West region of Cameroon: a cross-sectional study. BMC Health Serv Res. 2025 Oct 3;25(1):1303. doi: 10.1186/s12913-025-13467-1. PMID 41044580